CLINICAL TRIAL: NCT04235348
Title: The Impact of Red Meat and Whole-grains Intake on the Colonic Mucus' Thickness, Colonic MUC-2 Expression Rate and the Inflammatory Markers in the Blood.
Brief Title: The Impact of Red Meat and Whole-grains Intake on the Colonic Mucosal Barrier
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Horizon 2020 - European Commission (Other); Hospital of Southern Jutland (Other); Knud and Edith Eriksens fond (Unknown)
Responsible Party: Sponsor
Other Study IDs: ColonicMucus
Record Dates: First submitted 2019-12-10; First posted 2020-01-21 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-12

CONDITIONS: Mucus Colitis; Inflammation, Colon; Dietary Exposure
Keywords: Colonic mucus; Mucosal barrier; Red meat; Whole grain; Dietary fibers; Inflammation; Muc-2
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Fecal samples in DNA- stabilizing medium
  * Biopsies from the colon sigmoideum immediately frozen in nitrogen liquid
  * Biopsies from the colon sigmoideum in RNAlater, and frozen under -80 degree celsius
  * Blood samples
  * Spot-urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BELIEVE: Consists of subjects referred to a colonoscopy between June 1, 2017, and December 1, 2019, in the hospital of Southern Denmark

SUMMARY:
This study evaluates the impact of red meat and whole-grain intake on the colonic mucosal barrier and the dietary impact of these groups on the induced low-grade inflammation

DETAILED DESCRIPTION:
The mucus layer in the colon is a continuous barrier separating the epithelial cells from faecal enzymes, bacteria, toxic and other components. The colonic mucus layer in patients with Crohn's Disease and Ulcerative Colitis was previously demonstrated to be thinner and more permeable compared to healthy subjects.

The colonic mucus is composed of glycoproteins held together trough unstable disulfide bridges. The digestion of red meat is associated with monosulfide production, which could bind to the disulfide molecules, make more stable trisulfide molecules, and thus destroy the mucus architecture. Moreover, different bacteria were previously linked to red meat intake and were associated with a degradation of the colonic mucus such as akkermansia muciniphila.

From the other side, the fermentation of the undigested fibres, primarily in whole-grains, is associated with the production of short-chain fatty acids, which was related to a local anti-inflammatory effect.

In this study, we hypothesise:

1. High consumption of red meat is associated with a thinner colonic mucus layer;
2. High consumption of whole-grain fibres is associated with a thicker colonic mucus layer;
3. Mucin-2 gene expression is different between patients with high red meat consumption vs low red meat consumption;
4. Mucin-2 gene expression is different between patients with high whole-grain consumption vs low whole-grain intake;
5. The level of inflammatory markers in blood "IL-1beta, IL-4, IL-6, IL-10, Hs-CRP, and TNF-alfa is higher in subjects with high red meat and low whole-grain intake.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to a colonoscopy in the Hospital of Southern Denmark
* Subjects able to read and understand Danish
* Mentally habile subjects
* Subjects who accept to be a part of the project

Exclusion Criteria:

* History of active cancer
* A recent colonoscopy (less than 3 months ago )
* Anamnesis of Inflammatory bowel diseases.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects referred to a colonoscopy in the Hospital of Southern Denmark, and who met the eligibility criteria of this study were included.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Colonic mucus thickness | November 30,2019
  We will evaluate the thickness of the inner mucus layer in 38 biopsies of subjects, at the upper and lower quartiles of red meat and whole-grain consumption

SECONDARY OUTCOMES:
Muc-2 gene expression | December 10, 2019
  Using real time PCR, we will examine the association between the expression of mucin 2 gene in relation to red meat and whole grain fiber intake
Inflammatory markers in blood (IL-1beta, IL-4, IL-6, IL-10, Hs-CRP, and TNF-alfa) | January 1-2020
  These markers will be evaluated in relation to red meat and whole-grain intake

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Jawhara, M.D., Principal Investigator — The University of Southern Denmark
Locations (1):
- Hospital og Southern Jutland, Aabenraa, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jawhara M, Sorensen SB, Heitmann BL, Halldorsson ThornI, Pedersen AK, Andersen V. The Relation between Red Meat and Whole-Grain Intake and the Colonic Mucosal Barrier: A Cross-Sectional Study. Nutrients. 2020 Jun 12;12(6):1765. doi: 10.3390/nu12061765. PMID 32545531